CLINICAL TRIAL: NCT03258632
Title: Improving Outcomes Among Medical/Surgical Inpatients With Alcohol Use Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 15-298
Record Dates: First submitted 2017-08-15; First posted 2017-08-23 (Actual); Results first posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (No Intervention): Under usual care, when a patient screens positive on the AUDIT-C administered at intake, a provider (social worker, nurse) provides Brief Intervention (BI), i.e., tells the patient that problems are associated with alcohol use, and about recommended drinking limits; notes the patient as ready to change drinking or not, and as agreeing to treatment or not. If the patient agrees to treatment, specialty addiction services are notified.
- Intervention (Experimental): Patients will attend one 50-minute individual session with a Decision Coach (a trained clinical provider, e.g., MSW). Patients in DO-MoST will also attend 6 biweekly 15-minute telephone sessions from the same Decision Coach.
  Interventions: Behavioral: Drinking Options - Motivate, Shared Decisions, Telemonitor (DO-MoST)

INTERVENTIONS:
Behavioral: Drinking Options - Motivate, Shared Decisions, Telemonitor (DO-MoST) — Patients will attend one 50-minute individual session with a Decision Coach (a trained clinical provider, e.g., MSW). Patients in DO-MoST will also attend 6 biweekly 15-minute telephone sessions from the same Decision Coach.
  Arms: Intervention

SUMMARY:
This project aims to help Veterans who are in medical treatment and have untreated alcohol problems. First, the investigators adapted a Decision Aid that explains alcohol-related treatment options and their risks and benefits. Then, the investigators are determining the effectiveness of an intervention called DO-MoST (for Drinking Options-Motivate, Shared Decisions, Telemonitor), whereby a Decision Coach helps Veterans make decisions about alcohol-related behaviors and treatments they prefer, and keeps in contact by phone to continue to help with drinking and treatment decisions. DO-MoST is designed to increase rates at which Veterans decide to reduce or quit drinking, and begin and remain in treatment, and to improve drinking- and medical-related outcomes over time. It may also decrease Veterans' use of expensive health services such as hospitalizations and emergency visits. Finally, the investigators will study how VA can use DO-MoST on an ongoing, more widespread basis. The project should increase patient-centered health care for Veterans with alcohol problems to benefit their recovery.

DETAILED DESCRIPTION:
In fiscal year 2014, over 57,000 Veterans with diagnosed alcohol use disorders (AUDs) received VHA inpatient medical-surgical services. This likely underrepresents the prevalence of AUDs among Veteran inpatients, because these conditions often go undiagnosed during hospital stays. The high prevalence of AUDs among VHA medical and surgical patients is of critical concern because AUDs and medical conditions exacerbate one another, and their co-occurrence increases the use of costly health services. Yet, there are no evidence-based strategies that improve outcomes in this patient population by means of increased utilization (initiation, engagement) of AUD treatment services. The investigators have identified Drinking Options: Motivate, Shared Decisions, Telemonitor (DO-MoST) as a potential solution to the critical need for evidence-based strategies.

This project is evaluating DO-MoST as a new and innovative intervention to facilitate the transition from medical-surgical care to AUD treatment in primary and specialty care settings, thereby improving Veterans' AUD and medical outcomes. DO-MoST entails use of motivational interviewing and a decision aid during the inpatient stay to facilitate informed choices about drinking options and resources for help to change drinking, if desired, followed by telephone calls with the patient to continue to motivate and support decisions. In addition to determining the effectiveness of DO-MoST, this project includes a process evaluation - that is, will gather information from providers and patients on DO-MoST's implementation at the two project sites - to inform VA's potential widespread implementation of DO-MoST with medical-surgical patients with AUDs.

Using an effectiveness/implementation Hybrid Type 1 design, incorporating a randomized controlled trial (RCT) and process evaluation to facilitate future implementation, this project has three Specific Aims.

Aim 1: Adapt a decision aid being implemented with AUD patients in non-VA primary care settings to be appropriate for Veterans with AUDs in medical-surgical treatment settings. With this prototype, the investigators will conduct alpha testing with patients and providers, and adapt and pilot the decision aid to finalize it for use in the RCT.

Aim 2: Conduct DO-MoST at two VA facilities (Ann Arbor and Palo Alto) and evaluate its effectiveness.

The primary hypotheses are: Patients in DO-MoST, compared to patients in usual care (UC), will be more likely to (1) utilize AUD help (initiate, engage), (2) have better AUD (fewer heavy drinking days) and medical (physical status) outcomes, and (3) have fewer and more delayed acute care episodes (Emergency Department visits, rehospitalizations). Patients will be assessed at baseline, and 3, 6, and 12 months post-baseline, for outcomes and non-VA health care; VA health care will be assessed with VA databases. GLMM analyses will be conducted to compare the UC and DO-MoST groups on course of outcomes.

Aim 3: Conduct a qualitative process evaluation to inform the wider implementation of DO-MoST, using the RE-AIM (Reach, Effectiveness, Adoption, Implementation, Maintenance) framework. The purpose is to provide guidance for VA facilities' broader adoption of DO-MoST in the future, including its possible adaptation for diverse subpopulations of Veterans, such as patients with mental health diagnoses (e.g., PTSD).

In summary, this project will develop a decision aid and comprehensively examine DO-MoST as a novel and groundbreaking approach to providing a bridge between medical-surgical treatment and AUD treatment. Decision Aids have been used successfully in a number of contexts, but never with medical-AUD patients. The investigator's operations partners from VHA Office of Mental Health and Suicide Prevention, and Medical Service, are committed to directly addressing the dangerous, costly pattern of Veterans obtaining medical-surgical services but not receiving the AUD treatment they need. The project is focused on priorities in the VA Blueprint for Excellence, of HSR&D Service, and of the PIs' HSR&D Centers of Innovation.

ELIGIBILITY:
Inclusion Criteria:

Medical-surgical inpatients with alcohol use disorder at the Ann Arbor or Palo Alto VA. Specifically:

* in a current episode of medical-surgical care,
* meet DSM 5 criteria for an AUD
* no specialty addiction treatment or weekly mutual-help group attendance within 60 days prior to the inpatient episode,
* no restricted access due to infection control requirements (e.g., TB, MRSA, C. diff),
* no significant cognitive impairment,
* ongoing access to a cell or land line telephone,
* at least one contact who will continue to know the patient's contact information, and (8) not having participated in an interview for Aim 1 of this project.

Exclusion Criteria:

See inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-12-26 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Timko, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (2):
- United States (2):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Timko C, Lewis M, Lor MC, Aldaco-Revilla L, Blonigen D, Ilgen M. Hazardous Drinking Interventions Delivered During Medical-Surgical Care: Patient and Provider Views. J Clin Psychol Med Settings. 2024 Mar;31(1):224-235. doi: 10.1007/s10880-023-09954-4. Epub 2023 Mar 23. PMID 36959430

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | Intervention
Started | 82 | 73
Completed | 70 | 60
Not Completed | 12 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Intervention | Total
Number analyzed (Participants) | 82 | 73 | 155
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 45 | 92
  >=65 years | 35 | 28 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (14.7) | 59.5 (12.6) | 59.4 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 76 | 67 | 143
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 5 | 5
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 10 | 6 | 16
  White | 49 | 49 | 98
  More than one race | 10 | 11 | 21
  Unknown or Not Reported | 9 | 2 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 82 | 73 | 155

OUTCOME MEASURES:

1. Primary Outcome: Time Line Follow Back
Description: The investigators will use the Timeline Follow-Back (TLFB) to assess abstinence from alcohol use during the 30 days preceding assessment. The TLFB is a widely used, standardized, calendar-based retrospective self-report assessment to quantify daily alcohol use. The investigators will examine the primary outcome of abstinence from alcohol use at 12-month follow-up.
Time Frame: Alcohol use in the past 30 days, assessed at 12-month follow-up
Population: Participants who completed follow-up.
Measure: Number; unit: percentage of participants abstinent
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 66 | 60
percentage of participants abstinent | 48 | 56
Statistical Analysis 1: Comparison: Usual Care vs Intervention; Test type: Superiority; p < .05, Mixed Models Analysis; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.73 to 1.90]

2. Secondary Outcome: Utilization of Substance Use-related Care
Description: The investigators used a TLFB approach to assess utilization of substance use-related care (any receipt of outpatient and/or residential treatment for alcohol and/or drug problems, yes or no) between baseline and the 12-month follow-up.
Time Frame: 12 months
Population: Consented participants
Measure: Count of Participants; unit: Participants
Groups:
- Usual Care: Randomly assigned to usual care
- Intervention: Randomly assigned to DO-MoST
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 66 | 60
Participants | 21 | 6

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of study entry until the end of planned study participation which was 12 months.
Arm/Group | Usual Care | Intervention
All-Cause Mortality (participants affected / at risk) | 5/82 | 3/73
Serious Adverse Events (participants affected / at risk) | 19/82 | 10/73
Other Adverse Events (participants affected / at risk) | 0/82 | 0/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=82) | Intervention (N=73)
Hospitalization (Surgical and medical procedures) | 19 (19) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT03258632/Prot_SAP_000.pdf